CLINICAL TRIAL: NCT04660409
Title: Assessment of the Correlation Between Serum Levels of Adropin and Degree of Severity of Chronic Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Yotam Kolben, Principle Investigator, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ADROPINHCC- HMO-CTIL
Record Dates: First submitted 2020-11-24; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Chronic Liver Disease and Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Child Pugh A (Other)
  Interventions: Diagnostic Test: Blood test for serum Adropin
- Child Pugh B (Other)
  Interventions: Diagnostic Test: Blood test for serum Adropin
- Child Pugh C (Other)
  Interventions: Diagnostic Test: Blood test for serum Adropin
- HCC (Other)
  Interventions: Diagnostic Test: Blood test for serum Adropin
- Healthy (Other)
  Interventions: Diagnostic Test: Blood test for serum Adropin

INTERVENTIONS:
Diagnostic Test: Blood test for serum Adropin — Blood test for serum Adropin

SUMMARY:
Injury to the liver parenchyma associated with an influx of acute or chronic inflammatory cells is termed hepatitis. Cirrhosis refers to a progressive, diffuse, fibrosing, nodular condition that disrupts the entire normal architecture of the liver. Patients with chronic liver disease have sustained hepatic inflammation, fibrosis, and aberrant hepatocyte regeneration. These abnormalities can cause cirrhosis and favor a series of genetic and epigenetic events that culminate in the formation of dysplastic nodules, which are actually preneoplastic lesions . Hepatocellular carcinoma can also arise in patients who have chronic liver disease but does not have established cirrhosis or marked inflammation.

The "gold standard" for evaluation and follow up of liver fibrosis and cirrhosis is liver biopsy. It's a costly procedure with risks of severe complications, with sampling error and problematic long term follow up. Non-invasive tools are broadly used with good results, but none of the commonly used methods is perfect. In one meta-analysis, different methods were compared for diagnosis of cirrhosis in Non-alcoholic fatty liver disease (NAFLD) patients. For example (sensitivity; specificity): APRI (56.2% ;83.6%), FibroScan M Probe (78.2%; 90.8%), MRE (86.6%; 93.4%) . Child-Pugh classification and model for end-stage liver disease (MELD) scores are used as measures for assessment of degree of severity of liver disease. These models have some drawbacks; Ascites and encephalopathy included in Child-Pugh classification are subjective and may be variable according to the physician's judgment and the use of diuretics and lactulose. INR which appears in both methods does not sufficiently reflect coagulopathy and liver function and is also variable throughout different laboratories. Both are not sensitive enough for short interval periods.

One of the major complications of cirrhosis and chronic hepatitis is Hepatocellular carcinoma (HCC). Most guidelines recommend cirrhotic patients to undergo abdominal ultrasound every 6 much to detect HCC, given the expected tumor growth rate in the target population. Although widely use, the combination of ultrasound (US) with Alpha fetoprotein (AFP) is not recommended for surveillance in patients with active liver inflammation as the 6-8% gain in the detection rate does not counterbalance the increase in false positive results. Like in previous issues, a specific, cost effective marker is still needed.

Adropin is a 76-amino-acids secreted peptide, which is encoded by the Enho gene. The exact physiological role of Adropin in the liver is unknown. However, high levels of Adropin are correlated with low incidence of Type 2 Diabetes Mellitus, higher levels of HDL cholesterol, lower body-mass index (BMI), LDL cholesterol, Triglyceride levels and blood pressure.

Obesity has been recognized long ago as a significant risk factor for developing cancer and is an independent risk factor for HCC in patients with alcoholic (odds ratio 3.2) and cryptogenic (odds ratio 11.1) cirrhosis Serum Adropin levels were decreased and negatively correlated with liver injury in non-alcoholic steatohepatitis (NASH) mice. Knockout of Adropin significantly exacerbated hepatic steatosis, inflammatory responses and fibrosis in mice. Furthermore, the treatment with Adropin bioactive peptides slowed NASH progression in mice.

In search for a good diagnostic and prognostic marker in patients with liver disease, Adropin should be further investigated in humans.

In this Open-label, single-center study, 50 adults (>18) male and female with any degree of chronic liver disease will undergo a single blood test for serum levels of Adropin. Levels will be measured using ELISA technique. The results will be compared with the Child Pugh and MELD scores, liver enzymes, lipid profile, coagulation factors and fibroscan results based on the patients' clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 18 Years to 80 Years (Adult) Sexes Eligible for Study: All

  1. Diagnosis of chronic liver disease of any etiology.
  2. Females of childbearing potential must be non-pregnant
  3. No known history of significant neurological, renal, cardiovascular, respiratory (asthma), endocrinological, gastrointestinal, primary hematopoietic disease, neoplasm, or any other clinically significant medical disorder other than liver disease and the metabolic syndrome in patients with NASH.
  4. Patients must satisfy a medical examiner about their fitness to participate in the study.
  5. Patients must provide written informed consent to participate in the study.

Exclusion Criteria:

- 1. Patients with evidence of other serious infectious, autoimmune, hepatic, nephritic or systemic disease or compromised organ function except for the metabolic syndrome in patients with NASH.

2. Patients with any acute medical situation (e.g. acute infection) within 48 hours of blood tests.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
correlation between degree of severity of chronic liver disease and serum adropin levels. | 1 year
  correlation between degree of severity of chronic liver disease and serum adropin levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah medical center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No